CLINICAL TRIAL: NCT05923112
Title: BESPONSA® INJECTION 1 MG SPECIAL INVESTIGATION
Brief Title: BESPONSA Injection 1 mg Special Investigation
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1931024; NCT05923112 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Acute Lymphocytic Leukemia
Keywords: Drug use investigation in Japan
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to learn about the safety and effectiveness of BESPONSA. BESPONSA is approved for treatment of relapsed or refractory CD22-positive acute lymphocytic leukemia.

Registration criteria for this study is all patients who starting BESPONSA in Japan from its launch to the market to April 30, 2020.

All patients in this study will receive BESPONSA according to the prescriptions.

Patients will be followed up as follow.

* 52 weeks for patients who did not have a HSCT (Hematopoietic Stem Cell Transplant) within 52 weeks after starting BESPONSA.
* Up to 52 weeks after a HSCT for patients who had a HSCT within 52 weeks after starting BESPONSA.

ELIGIBILITY:
Inclusion Criteria:

* All patients prescribed BESPONSA

Exclusion Criteria:

* None

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who received BESPONSA
Sampling Method: Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1931024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 421 participants were considered to be enrolled because they used this drug after marketing. CRFs were collected from 383 of these participants. Although data were analyzed from 383 participants for all-case surveillance, only 136 participants provided informed consent for results disclosure and are reported in the record.
Groups:
- BESPONSA Injection 1mg (Inotuzumab Ozogamicin): Participants who received BESPONSA Injection 1mg as indicated in the approved local product document were observed for up to 104 weeks. The dosage can be adjusted as per physician's discretion. The observation period was divided into two phases: the treatment phase and the follow-up phase. The treatment phase was from the first day of treatment to 28 days after the last treatment, and safety was observed for adverse events, and effectiveness was observed for hematological response and overall survival (OS). The follow-up phase was from the 29th day after the last administration to week 52 for participants who did not undergo hematopoietic stem cell transplant (HSCT) within 52 weeks of the start of administration, or was up to 52 weeks after HSCT for participants who underwent HSCT within 52 weeks of the start of administration. Safety was observed for venoocclusive disease (VOD)/sinusoidal obstruction syndrome (SOS), and effectiveness was observed as survival time.
Period: Overall Study
Arm/Group | BESPONSA Injection 1mg (Inotuzumab Ozogamicin)
Started | 383
Completed | 136
Not Completed | 247
Not completed — Protocol Violation | 4
Not completed — No informed consent on publication of study results | 243

BASELINE CHARACTERISTICS:
Population: 383 participants contributed to the all-case surveillance analysis, regardless of whether they consented to disclosure of results. 247 participants were excluded from the safety analysis set due to the following: protocol violation (4 participants) and no informed consent on publication of study results (243 participants). 136 participants who provided consent for results disclosure completed the study. Overall, the safety analysis set comprised of 136 participants.
Groups:
- BESPONSA Injection 1mg (Inotuzumab Ozogamicin): Participants who received BESPONSA Injection 1mg as indicated in the approved local product document were observed for up to 104 weeks. The dosage can be adjusted as per physician's discretion. The observation period was divided into two phases: the treatment phase and the follow-up phase. The treatment phase was from the first day of treatment to 28 days after the last treatment, and safety was observed for adverse events, and effectiveness was observed for hematological response and OS. The follow-up phase was from the 29th day after the last administration to week 52 for participants who did not undergo HSCT within 52 weeks of the start of administration, or was up to 52 weeks after HSCT for participants who underwent HSCT within 52 weeks of the start of administration. Safety was observed for VOD/SOS, and effectiveness was observed as survival time.
Arm/Group | BESPONSA Injection 1mg (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 136
Age, Customized [Number; unit: participants]
  <15 years | 11
  ≥15 and <65 years | 61
  ≥65 years | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 67
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Adverse Drug Reactions
Description: An adverse drug reaction (ADR) was a treatment-related adverse event, and any untoward medical occurrence attributed to BESPONSA Injection 1mg in a participant who received BESPONSA Injection 1mg. A serious adverse drug reaction (SADR) was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: results in death; is life-threatening; requires inpatient hospitalization or prolongation of hospitalization; results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); results in congenital anomaly/birth defect.
Time Frame: From first dose up to 28 days after last dose. VOD/SOS: No HSCT: up to 52 weeks, HSCT: up to 104 weeks
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received BESPONSA Injection 1mg at least once. Participants with protocol violation and without informed consent on publication of study results were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | BESPONSA Injection 1mg (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 136
Participants
  ADR | 72
  SADR | 21

2. Primary Outcome: The Incidence of Liver Disorder Including VOD/SOS (ADRs)/ (All CTCAE Grades)
Description: Risk ratios for the proportion of participants with ADRs in different subgroups were determined. However, if there was a category with fewer than 10 participants and it was considered difficult to determine the risk ratio for that category after reconsideration, the risk ratio was not determined for that category.
  ADRs meeting definition of liver disorder including safety specification events of VOD/SOS were analyzed by each of the following factors: Age; Hepatic impairment; Medical history (past) - VOD/SOS, Hepatitis or hepatic disease; Medical history (present) - VOD/SOS, Hepatitis or hepatic disease; Eastern Cooperative Oncology Group performance status (ECOG PS); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels; gamma glutamyl transpeptidase (γ-GTP) level; Total bilirubin level; Platelet count; Peripheral blast count; Salvage line of the induction treatment with this drug; HSCT before the start of this drug.
Time Frame: No HSCT: up to 52 weeks, HSCT: up to 104 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BESPONSA Injection 1mg (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 136
Participants | 25
Statistical Analysis 1: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 15 years, ≥ 15 to < 65 years]; Test type: Other — Estimation; Risk Ratio (RR) = 1.008, 95% CI 2-sided [0.258 to 3.940] — Risk Ratio of age "< 15 years" to "≥ 15 to < 65 years"
Statistical Analysis 2: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 65 years, ≥ 15 to < 65 years]; Test type: Other — Estimation; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.497 to 2.177] — Risk Ratio of age "≥ 65 years" to "≥ 15 to < 65 years"
Statistical Analysis 3: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 18 years, ≥ 18 to < 55 years]; Test type: Other — Estimation; Risk Ratio (RR) = 1.084, 95% CI 2-sided [0.317 to 3.710] — Risk Ratio of age "< 18 years" to "≥ 18 to < 55 years"
Statistical Analysis 4: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 55 years, ≥ 18 to < 55 years]; Test type: Other — Estimation; Risk Ratio (RR) = 1.212, 95% CI 2-sided [0.536 to 2.740] — Risk Ratio of age "≥ 55 years" to "≥ 18 to < 55 years"
Statistical Analysis 5: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 15 years, ≥ 15 to < 40 years]; Test type: Other — Estimation; Risk Ratio (RR) = 1.091, 95% CI 2-sided [0.247 to 4.827] — Risk Ratio of age "< 15 years" to "≥ 15 to < 40 years"
Statistical Analysis 6: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 40 years, ≥ 15 to < 40 years]; Test type: Other — Estimation; Risk Ratio (RR) = 1.137, 95% CI 2-sided [0.461 to 2.801] — Risk Ratio of age "≥ 40 years" to "≥ 15 to < 40 years"
Statistical Analysis 7: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of hepatic impairment; Test type: Other — Estimation; Risk Ratio (RR) = 1.409, 95% CI 2-sided [0.493 to 4.030] — Risk Ratio of hepatic impairment "present" to "absent"
Statistical Analysis 8: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of past medical history - Hepatitis or hepatic disease; Test type: Other — Estimation; Risk Ratio (RR) = 1.096, 95% CI 2-sided [0.301 to 3.994] — Risk Ratio of past medical history - Hepatitis or hepatic disease "present" to "absent"
Statistical Analysis 9: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of present medical history - Hepatitis or hepatic disease; Test type: Other — Estimation; Risk Ratio (RR) = 1.409, 95% CI 2-sided [0.493 to 4.030] — Risk Ratio of present medical history - Hepatitis or hepatic disease "present" to "absent"
Statistical Analysis 10: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 2.954, 95% CI 2-sided [1.172 to 7.445] — Risk Ratio of ECOG PS before the start of this drug "0" to "1"
Statistical Analysis 11: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 1.152, 95% CI 2-sided [0.299 to 4.432] — Risk Ratio of ECOG PS before the start of this drug "≥ 2" to "1"
Statistical Analysis 12: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.873, 95% CI 2-sided [0.113 to 6.743] — Risk Ratio of ECOG PS before the start of this drug "not performed" to "1"
Statistical Analysis 13: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of AST and ALT levels immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 1.158, 95% CI 2-sided [0.545 to 2.461] — Risk Ratio of AST and ALT levels immediately before the start of this drug "either > 1.5 × the institutional upper limit normal range (IULN)" to "≤ 1.5 × IULN"
Statistical Analysis 14: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of γ-GTP level immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.59, 95% CI 2-sided [0.280 to 1.244] — Risk Ratio of γ-GTP level immediately before the start of this drug "> 50 IU/L" to "≤ 50 IU/L"
Statistical Analysis 15: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of γ-GTP level immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.267, 95% CI 2-sided [0.038 to 1.862] — Risk Ratio of γ-GTP level immediately before the start of this drug "not performed" to "≤ 50 IU/L"
Statistical Analysis 16: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of platelet count immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.413, 95% CI 2-sided [0.201 to 0.849] — Risk Ratio of platelet count immediately before the start of this drug "< 10 × 10⁴/μL" to "≥ 10 × 10⁴/μL"
Statistical Analysis 17: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of peripheral blast count immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.299, 95% CI 2-sided [0.075 to 1.194] — Risk Ratio of peripheral blast count immediately before the start of this drug "> 1000 /μL" to "≤ 1000 /μL"
Statistical Analysis 18: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of salvage line of the induction treatment with this drug; Test type: Other — Estimation; Risk Ratio (RR) = 2.415, 95% CI 2-sided [0.917 to 6.362] — Risk Ratio of salvage line of the induction treatment with this drug "2nd" to "1st"
Statistical Analysis 19: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of salvage line of the induction treatment with this drug; Test type: Other — Estimation; Risk Ratio (RR) = 1.688, 95% CI 2-sided [0.612 to 4.655] — Risk Ratio of salvage line of the induction treatment with this drug "3rd or later" to "1st"
Statistical Analysis 20: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of HSCT before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.901, 95% CI 2-sided [0.408 to 1.990] — Risk Ratio of HSCT before the start of this drug "performed" to "not performed"

3. Primary Outcome: The Incidence of Liver Disorder Including VOD/SOS (ADRs)/ (CTCAE Grade 3 or Higher)
Description: Risk ratios for the proportion of participants with ADRs in different subgroups was determined. However, if there was a category with fewer than 10 participants and it was considered difficult to determine the risk ratio for that category after reconsideration, the risk ratio was not determined for that category. In category(A) The risk ratio was calculable; however, the confidence interval could not be estimated due to the absence of ADRs in the numerator.
  ADRs meeting definition of liver disorder including safety specification events of VOD/SOS were analyzed by each of the following factors: Age; Hepatic impairment; Medical history (past) - VOD/SOS, Hepatitis or hepatic disease; Medical history (present) - VOD/SOS, Hepatitis or hepatic disease; ECOG PS; AST and ALT levels; γ-GTP level; Total bilirubin level; Platelet count; Peripheral blast count; Salvage line of the induction treatment with this drug; HSCT before the start of this drug.
Time Frame: No HSCT: up to 52 weeks, HSCT: up to 104 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BESPONSA Injection 1mg (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 136
Participants | 15
Statistical Analysis 1: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 15 years, ≥ 15 to < 65 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0.616, 95% CI 2-sided [0.086 to 4.391] — Risk Ratio of age "< 15 years" to "≥ 15 to < 65 years"
Statistical Analysis 2: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 65 years, ≥ 15 to < 65 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0.53, 95% CI 2-sided [0.188 to 1.491] — Risk Ratio of age "≥ 65 years" to "≥ 15 to < 65 years"
Statistical Analysis 3: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 18 years, ≥ 18 to < 55 years]; Test type: Other — Estimation; Risk Ratio (RR) = 1.012, 95% CI 2-sided [0.217 to 4.723] — Risk Ratio of age "< 18 years" to "≥ 18 to < 55 years"
Statistical Analysis 4: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 55 years, ≥ 18 to < 55 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0.905, 95% CI 2-sided [0.316 to 2.594] — Risk Ratio of age "≥ 55 years" to "≥ 18 to < 55 years"
Statistical Analysis 5: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 15 years, ≥ 15 to < 40 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0.682, 95% CI 2-sided [0.085 to 5.455] — Risk Ratio of age "< 15 years" to "≥ 15 to < 40 years"
Statistical Analysis 6: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 40 years, ≥ 15 to < 40 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0.789, 95% CI 2-sided [0.267 to 2.335] — Risk Ratio of age "≥ 40 years" to "≥ 15 to < 40 years"
Statistical Analysis 7: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of hepatic impairment; Test type: Other — Estimation; Risk Ratio (RR) = 2.583, 95% CI 2-sided [0.845 to 7.900] — Risk Ratio of hepatic impairment "present" to "absent"
Statistical Analysis 8: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of past medical history - Hepatitis or hepatic disease; Test type: Other — Estimation; Risk Ratio (RR) = 0.9, 95% CI 2-sided [0.131 to 6.163] — Risk Ratio of past medical history - Hepatitis or hepatic disease "present" to "absent"
Statistical Analysis 9: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of present medical history - Hepatitis or hepatic disease; Test type: Other — Estimation; Risk Ratio (RR) = 2.583, 95% CI 2-sided [0.845 to 7.900] — Risk Ratio of present medical history - Hepatitis or hepatic disease "present" to "absent"
Statistical Analysis 10: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 2.769, 95% CI 2-sided [0.796 to 9.630] — Risk Ratio of ECOG PS before the start of this drug "0" to "1"
Statistical Analysis 11: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 1.92, 95% CI 2-sided [0.418 to 8.827] — Risk Ratio of ECOG PS before the start of this drug "≥ 2" to "1"
Statistical Analysis 12: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0 — The risk ratio was reported as participants in this group are related to Category(A); Regarding Risk Ratio of ECOG PS before the start of this drug "not performed" to "1"
Statistical Analysis 13: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of AST and ALT levels immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.615, 95% CI 2-sided [0.184 to 2.062] — Risk Ratio of AST and ALT levels immediately before the start of this drug "either > 1.5 × the institutional upper limit normal range (IULN)" to "≤ 1.5 ×IULN"
Statistical Analysis 14: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of γ-GTP level immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.656, 95% CI 2-sided [0.249 to 1.729] — Risk Ratio of γ-GTP level immediately before the start of this drug "> 50 IU/L" to "≤ 50 IU/L"
Statistical Analysis 15: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of γ-GTP level immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0 — The risk ratio was reported as participants in this group are related to Category(A); Regarding Risk Ratio of γ-GTP level immediately before the start of this drug "not performed" to "≤ 50 IU/L"
Statistical Analysis 16: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of platelet count immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.707, 95% CI 2-sided [0.273 to 1.836] — Risk Ratio of platelet count immediately before the start of this drug "< 10 × 10⁴/μL" to "≥ 10 × 10⁴/μL"
Statistical Analysis 17: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of peripheral blast count immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.245, 95% CI 2-sided [0.034 to 1.790] — Risk Ratio of peripheral blast count immediately before the start of this drug "> 1000 /μL" to "≤ 1000 /μL"
Statistical Analysis 18: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of salvage line of the induction treatment with this drug; Test type: Other — Estimation; Risk Ratio (RR) = 2.927, 95% CI 2-sided [0.832 to 10.294] — Risk Ratio of salvage line of the induction treatment with this drug "2nd" to "1st"
Statistical Analysis 19: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of salvage line of the induction treatment with this drug; Test type: Other — Estimation; Risk Ratio (RR) = 1.25, 95% CI 2-sided [0.296 to 5.279] — Risk Ratio of salvage line of the induction treatment with this drug "3rd or later" to "1st"
Statistical Analysis 20: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of HSCT before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 1.545, 95% CI 2-sided [0.588 to 4.058] — Risk Ratio of HSCT before the start of this drug "performed" to "not performed"

4. Primary Outcome: The Incidence of Myelosuppression (ADRs)/ (All CTCAE Grades)
Description: Risk ratios for the proportion of participants with ADRs in different subgroups was determined. However, if there was a category with fewer than 10 participants and it was considered difficult to determine the risk ratio for that category after reconsideration, the risk ratio was not determined for that category.
  ADRs meeting definition of safety specification events of myelosuppression were analyzed by each of the following factors: Age; Hepatic impairment; Renal impairment; Total dose per cycle > 1.8 mg/m2; ECOG PS; White blood cell count; Neutrophil count; Platelet count; Salvage line of the induction treatment with this drug; HSCT before the start of this drug.
Time Frame: From the start date of administration to Day 28 post-final dose, approximately 27 weeks for HSCT and no HSCT participants
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BESPONSA Injection 1mg (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 136
Participants | 52
Statistical Analysis 1: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 15 years, ≥ 15 to < 65 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0.528, 95% CI 2-sided [0.144 to 1.939] — Risk Ratio of age "< 15 years" to "≥ 15 to < 65 years"
Statistical Analysis 2: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 65 years, ≥ 15 to < 65 years]; Test type: Other — Estimation; Risk Ratio (RR) = 1.316, 95% CI 2-sided [0.849 to 2.041] — Risk Ratio of age "≥ 65 years" to "≥ 15 to < 65 years"
Statistical Analysis 3: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 18 years, ≥ 18 to < 55 years]; Test type: Other — Estimation; Risk Ratio (RR) = 1.084, 95% CI 2-sided [0.500 to 2.351] — Risk Ratio of age "< 18 years" to "≥ 18 to < 55 years"
Statistical Analysis 4: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 55 years, ≥ 18 to < 55 years]; Test type: Other — Estimation; Risk Ratio (RR) = 1.293, 95% CI 2-sided [0.781 to 2.142] — Risk Ratio of age "≥ 55 years" to "≥ 18 to < 55 years"
Statistical Analysis 5: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 15 years, ≥ 15 to < 40 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0.455, 95% CI 2-sided [0.120 to 1.715] — Risk Ratio of age "< 15 years" to "≥ 15 to < 40 years"
Statistical Analysis 6: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 40 years, ≥ 15 to < 40 years]; Test type: Other — Estimation; Risk Ratio (RR) = 1, 95% CI 2-sided [0.605 to 1.653] — Risk Ratio of age "≥ 40 years" to "≥ 15 to < 40 years"
Statistical Analysis 7: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of hepatic impairment; Test type: Other — Estimation; Risk Ratio (RR) = 1.099, 95% CI 2-sided [0.542 to 2.228] — Risk Ratio of hepatic impairment "present" to "absent"
Statistical Analysis 8: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 1.069, 95% CI 2-sided [0.667 to 1.714] — Risk Ratio of ECOG PS before the start of this drug "0" to "1"
Statistical Analysis 9: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.909, 95% CI 2-sided [0.485 to 1.705] — Risk Ratio of ECOG PS before the start of this drug "≥ 2" to "1"
Statistical Analysis 10: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.459, 95% CI 2-sided [0.125 to 1.688] — Risk Ratio of ECOG PS before the start of this drug "not performed" to "1"
Statistical Analysis 11: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of white blood cell count immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.889, 95% CI 2-sided [0.580 to 1.362] — Risk Ratio of white blood cell count immediately before the start of this drug "≥ 4000/mm³" to "< 4000/mm³"
Statistical Analysis 12: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of neutrophil count immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 1.121, 95% CI 2-sided [0.728 to 1.725] — Risk Ratio of neutrophil count immediately before the start of this drug "≥ 2000/mm³" to "< 2000/mm³"
Statistical Analysis 13: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of platelet count immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.639 to 1.536] — Risk Ratio of platelet count immediately before the start of this drug "< 10 × 10⁴/μL" to "≥ 10 × 10⁴/μL"
Statistical Analysis 14: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of salvage line of the induction treatment with this drug; Test type: Other — Estimation; Risk Ratio (RR) = 1.996, 95% CI 2-sided [1.093 to 3.643] — Risk Ratio of salvage line of the induction treatment with this drug "2nd" to "1st"
Statistical Analysis 15: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of salvage line of the induction treatment with this drug; Test type: Other — Estimation; Risk Ratio (RR) = 1.79, 95% CI 2-sided [0.977 to 3.279] — Risk Ratio of salvage line of the induction treatment with this drug "3rd or later" to "1st"
Statistical Analysis 16: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of HSCT before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.772, 95% CI 2-sided [0.464 to 1.286] — Risk Ratio of HSCT before the start of this drug "performed" to "not performed"

5. Primary Outcome: The Incidence of Myelosuppression (ADRs)/ (CTCAE Grade 3 or Higher)
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BESPONSA Injection 1mg (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 136
Participants | 43
Statistical Analysis 1: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 15 years, ≥ 15 to < 65 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0.584, 95% CI 2-sided [0.158 to 2.159] — Risk Ratio of age "< 15 years" to "≥ 15 to < 65 years"
Statistical Analysis 2: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 65 years, ≥ 15 to < 65 years]; Test type: Other — Estimation; Risk Ratio (RR) = 1.104, 95% CI 2-sided [0.667 to 1.826] — Risk Ratio of age "≥ 65 years" to "≥ 15 to < 65 years"
Statistical Analysis 3: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 18 years, ≥ 18 to < 55 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0.973, 95% CI 2-sided [0.410 to 2.311] — Risk Ratio of age "< 18 years" to "≥ 18 to < 55 years"
Statistical Analysis 4: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 55 years, ≥ 18 to < 55 years]; Test type: Other — Estimation; Risk Ratio (RR) = 1.088, 95% CI 2-sided [0.624 to 1.897] — Risk Ratio of age "≥ 55 years" to "≥ 18 to < 55 years"
Statistical Analysis 5: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 15 years, ≥ 15 to < 40 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0.545, 95% CI 2-sided [0.141 to 2.108] — Risk Ratio of age "< 15 years" to "≥ 15 to < 40 years"
Statistical Analysis 6: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 40 years, ≥ 15 to < 40 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0.979, 95% CI 2-sided [0.547 to 1.753] — Risk Ratio of age "≥ 40 years" to "≥ 15 to < 40 years"
Statistical Analysis 7: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of hepatic impairment; Test type: Other — Estimation; Risk Ratio (RR) = 1.36, 95% CI 2-sided [0.662 to 2.793] — Risk Ratio of hepatic impairment "present" to "absent"
Statistical Analysis 8: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.769, 95% CI 2-sided [0.439 to 1.349] — Risk Ratio of ECOG PS before the start of this drug "0" to "1"
Statistical Analysis 9: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.507 to 1.816] — Risk Ratio of ECOG PS before the start of this drug "≥ 2" to "1"
Statistical Analysis 10: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.242, 95% CI 2-sided [0.036 to 1.627] — Risk Ratio of ECOG PS before the start of this drug "not performed" to "1"
Statistical Analysis 11: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of white blood cell count immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.848, 95% CI 2-sided [0.518 to 1.391] — Risk Ratio of white blood cell count immediately before the start of this drug "≥ 4000/mm³" to "< 4000/mm³"
Statistical Analysis 12: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of neutrophil count immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.945, 95% CI 2-sided [0.578 to 1.547] — Risk Ratio of neutrophil count immediately before the start of this drug "≥ 2000/mm³" to "< 2000/mm³"
Statistical Analysis 13: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of platelet count immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 1.156, 95% CI 2-sided [0.685 to 1.950] — Risk Ratio of platelet count immediately before the start of this drug "< 10 × 10⁴/μL" to "≥ 10 × 10⁴/μL"
Statistical Analysis 14: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of salvage line of the induction treatment with this drug; Test type: Other — Estimation; Risk Ratio (RR) = 2.195, 95% CI 2-sided [1.113 to 4.329] — Risk Ratio of salvage line of the induction treatment with this drug "2nd" to "1st"
Statistical Analysis 15: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of salvage line of the induction treatment with this drug; Test type: Other — Estimation; Risk Ratio (RR) = 1.667, 95% CI 2-sided [0.821 to 3.384] — Risk Ratio of salvage line of the induction treatment with this drug "3rd or later" to "1st"
Statistical Analysis 16: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of HSCT before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 1.004, 95% CI 2-sided [0.586 to 1.719] — Risk Ratio of HSCT before the start of this drug "performed" to "not performed"

6. Primary Outcome: The Incidence of Infections (ADRs)/ (All CTCAE Grades)
Description: Risk ratios for the proportion of participants with ADRs in different subgroups was determined. However, if there was a category with fewer than 10 participants and it was considered difficult to determine the risk ratio for that category after reconsideration, the risk ratio was not determined for that category. In category(A) The risk ratio was calculable; however, the confidence interval could not be estimated due to the absence of ADRs in the numerator. In category (B) The risk ratio and confidence interval could not be estimated because no ADRs were observed in either the numerator, the denominator, or both.
  ADRs meeting definition of safety specification events of infection were analyzed by each of the following factors: Age; Hepatic impairment; Renal impairment; Total dose per cycle > 1.8 mg/m2; ECOG PS; Salvage line of the induction treatment with this drug; HSCT before the start of this drug.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BESPONSA Injection 1mg (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 136
Participants | 7
Statistical Analysis 1: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 15 years, ≥ 15 to < 65 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0 — The risk ratio was reported as participants in this group are related to Category(A); Regarding Risk Ratio of age "< 15 years" to "≥ 15 to < 65 years"
Statistical Analysis 2: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 65 years, ≥ 15 to < 65 years]; Test type: Other — Estimation; Risk Ratio (RR) = 2.383, 95% CI 2-sided [0.480 to 11.824] — Risk Ratio of age "≥ 65 years" to "≥ 15 to < 65 years"
Statistical Analysis 3: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 18 years, ≥ 18 to < 55 years]; Test type: Other — Estimation; Risk Ratio (RR) = 2.529, 95% CI 2-sided [0.168 to 38.180] — Risk Ratio of age "< 18 years" to "≥ 18 to < 55 years"
Statistical Analysis 4: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 55 years, ≥ 18 to < 55 years]; Test type: Other — Estimation; Risk Ratio (RR) = 2.829, 95% CI 2-sided [0.342 to 23.432] — Risk Ratio of age "≥ 55 years" to "≥ 18 to < 55 years"
Statistical Analysis 5: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 15 years, ≥ 15 to < 40 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0 — The risk ratio was reported as participants in this group are related to Category(A); Regarding Risk Ratio of age "< 15 years" to "≥ 15 to < 40 years"
Statistical Analysis 6: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 40 years, ≥ 15 to < 40 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0.789, 95% CI 2-sided [0.161 to 3.862] — Risk Ratio of age "≥ 40 years" to "≥ 15 to < 40 years"
Statistical Analysis 7: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of hepatic impairment; Test type: Other — Estimation; Risk Ratio (RR) = 0 — The risk ratio was reported as participants in this group are related to Category(A); Regarding Risk Ratio of hepatic impairment "present" to "absent"
Statistical Analysis 8: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.923, 95% CI 2-sided [0.196 to 4.355] — Risk Ratio of ECOG PS before the start of this drug "0" to "1"
Statistical Analysis 9: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.64, 95% CI 2-sided [0.070 to 5.840] — Risk Ratio of ECOG PS before the start of this drug "≥ 2" to "1"
Statistical Analysis 10: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0 — The risk ratio was reported as participants in this group are related to Category(A); Regarding Risk Ratio of ECOG PS before the start of this drug "not performed" to "1"
Statistical Analysis 11: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of HSCT before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.386, 95% CI 2-sided [0.048 to 3.107] — Risk Ratio of HSCT before the start of this drug "performed" to "not performed"
Statistical Analysis 12: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of salvage line of the induction treatment with this drug; Test type: Other — Estimation; Regarding Risk Ratio of salvage line of the induction treatment with this drug "2nd" to "1st", the risk ratio was reported as participants in this group are related to Category(B)
Statistical Analysis 13: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of salvage line of the induction treatment with this drug; Test type: Other — Estimation; Regarding Risk Ratio of salvage line of the induction treatment with this drug "3rd or later" to "1st", the risk ratio was reported as participants in this group are related to Category(B)

7. Primary Outcome: The Incidence of Infections (ADRs)/ (CTCAE Grade 3 or Higher)
Description: as for outcome 6
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BESPONSA Injection 1mg (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 136
Participants | 4
Statistical Analysis 1: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 15 years, ≥ 15 to < 65 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0 — The risk ratio was reported as participants in this group are related to Category(A); Regarding Risk Ratio of age "< 15 years" to "≥ 15 to < 65 years"
Statistical Analysis 2: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 65 years, ≥ 15 to < 65 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0.953, 95% CI 2-sided [0.139 to 6.556] — Risk Ratio of age "≥ 65 years" to "≥ 15 to < 65 years"
Statistical Analysis 3: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 18 years, ≥ 18 to < 55 years]; Test type: Other — Estimation; Risk Ratio (RR) = 2.529, 95% CI 2-sided [0.168 to 38.180] — Risk Ratio of age "< 18 years" to "≥ 18 to < 55 years"
Statistical Analysis 4: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 55 years, ≥ 18 to < 55 years]; Test type: Other — Estimation; Risk Ratio (RR) = 1.132, 95% CI 2-sided [0.106 to 12.119] — Risk Ratio of age "≥ 55 years" to "≥ 18 to < 55 years"
Statistical Analysis 5: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 15 years, ≥ 15 to < 40 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0 — The risk ratio was reported as participants in this group are related to Category(A); Regarding Risk Ratio of age "< 15 years" to "≥ 15 to < 40 years"
Statistical Analysis 6: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 40 years, ≥ 15 to < 40 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0.316, 95% CI 2-sided [0.046 to 2.146] — Risk Ratio of age "≥ 40 years" to "≥ 15 to < 40 years"
Statistical Analysis 7: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of hepatic impairment; Test type: Other — Estimation; Risk Ratio (RR) = 0 — The risk ratio was reported as participants in this group are related to Category(A); Regarding Risk Ratio of hepatic impairment "present" to "absent"
Statistical Analysis 8: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.462, 95% CI 2-sided [0.043 to 4.928] — Risk Ratio of ECOG PS before the start of this drug "0" to "1"
Statistical Analysis 9: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.091 to 10.079] — Risk Ratio of ECOG PS before the start of this drug "≥ 2" to "1"
Statistical Analysis 10: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0 — The risk ratio was reported as participants in this group are related to Category(A); Regarding Risk Ratio of ECOG PS before the start of this drug "not performed" to "1"
Statistical Analysis 11: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of HSCT before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.772, 95% CI 2-sided [0.083 to 7.207] — Risk Ratio of HSCT before the start of this drug "performed" to "not performed"
Statistical Analysis 12: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of salvage line of the induction treatment with this drug; Test type: Other — Estimation; [other analysis details as in outcome 6, analysis 12]
Statistical Analysis 13: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of salvage line of the induction treatment with this drug; Test type: Other — Estimation; [other analysis details as in outcome 6, analysis 13]

8. Primary Outcome: The Incidence of Hemorrhage (ADRs)/ (All CTCAE Grades)
Description: Risk ratios for the proportion of participants with ADRs in different subgroups was determined. However, if there was a category with fewer than 10 participants and it was considered difficult to determine the risk ratio for that category after reconsideration, the risk ratio was not determined for that category. In category(A) The risk ratio was calculable; however, the confidence interval could not be estimated due to the absence of ADRs in the numerator. In category (B) The risk ratio and confidence interval could not be estimated because no ADRs were observed in either the numerator, the denominator, or both.
  ADRs meeting definition of safety specification events of hemorrhage were analyzed by each of the following factors: Age; Hepatic impairment; Renal impairment; Total dose per cycle > 1.8 mg/m2; ECOG PS; Salvage line of the induction treatment with this drug; HSCT before the start of this drug.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BESPONSA Injection 1mg (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 136
Participants | 2
Statistical Analysis 1: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of hepatic impairment; Test type: Other — Estimation; Risk Ratio (RR) = 0 — The risk ratio was reported as participants in this group are related to Category(A); Regarding Risk Ratio of hepatic impairment "present" to "absent"
Statistical Analysis 2: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.923, 95% CI 2-sided [0.059 to 14.352] — Risk Ratio of ECOG PS before the start of this drug "0" to "1"
Statistical Analysis 3: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0 — The risk ratio was reported as participants in this group are related to Category(A); Regarding Risk Ratio of ECOG PS before the start of this drug "≥ 2" to "1"
Statistical Analysis 4: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0 — The risk ratio was reported as participants in this group are related to Category(A); Regarding Risk Ratio of ECOG PS before the start of this drug "not performed" to "1"
Statistical Analysis 5: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of HSCT before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0 — The risk ratio was reported as participants in this group are related to Category(A); Regarding Risk Ratio of HSCT before the start of this drug "performed" to "not performed"
Statistical Analysis 6: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 15 years, ≥ 15 to < 65 years]; Test type: Other — Estimation; Regarding Risk Ratio of age "< 15 years" to "≥ 15 to < 65 years", the risk ratio was reported as participants in this group are related to Category(B)
Statistical Analysis 7: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 65 years, ≥ 15 to < 65 years]; Test type: Other — Estimation; Regarding Risk Ratio of age "≥ 65 years" to "≥ 15 to < 65 years", the risk ratio was reported as participants in this group are related to Category(B)
Statistical Analysis 8: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 18 years, ≥ 18 to < 55 years]; Test type: Other — Estimation; Regarding Risk Ratio of age "< 18 years" to "≥ 18 to < 55 years", the risk ratio was reported as participants in this group are related to Category(B)
Statistical Analysis 9: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 55 years, ≥ 18 to < 55 years]; Test type: Other — Estimation; Regarding Risk Ratio of age "≥ 55 years" to "≥ 18 to < 55 years", the risk ratio was reported as participants in this group are related to Category(B)
Statistical Analysis 10: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 15 years, ≥ 15 to < 40 years]; Test type: Other — Estimation; Regarding Risk Ratio of age "< 15 years" to "≥ 15 to < 40 years", the risk ratio was reported as participants in this group are related to Category(B)
Statistical Analysis 11: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 40 years, ≥ 15 to < 40 years]; Test type: Other — Estimation; Regarding Risk Ratio of age "≥ 40 years" to "≥ 15 to < 40 years", the risk ratio was reported as participants in this group are related to Category(B)
Statistical Analysis 12: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of salvage line of the induction treatment with this drug; Test type: Other — Estimation; [other analysis details as in outcome 6, analysis 12]
Statistical Analysis 13: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of salvage line of the induction treatment with this drug; Test type: Other — Estimation; [other analysis details as in outcome 6, analysis 13]

9. Primary Outcome: The Incidence of Hemorrhage (ADRs)/ (CTCAE Grade 3 or Higher)
Description: Risk ratios for the proportion of participants with ADRs in different subgroups was determined. However, if there was a category with fewer than 10 participants and it was considered difficult to determine the risk ratio for that category after reconsideration, the risk ratio was not determined for that category.
  ADRs meeting definition of safety specification events of hemorrhage were analyzed by each of the following factors: Age; Hepatic impairment; Renal impairment; Total dose per cycle > 1.8 mg/m2; ECOG PS; Salvage line of the induction treatment with this drug; HSCT before the start of this drug.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BESPONSA Injection 1mg (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 136
Participants | 0

10. Primary Outcome: Early Death After HSCT
Description: Risk ratios for the proportion of participants with early death in different subgroups was determined. However, if there was a category with fewer than 10 participants and it was considered difficult to determine the risk ratio for that category after reconsideration, the risk ratio was not determined for that category.
  Participants in the safety analysis set who underwent HSCT after the start of BESPONSA Injection 1mg and have completed the study were included in the analysis. Early death after HSCT was defined as death occurring within 100 days after the first HSCT following the start of BESPONSA Injection 1mg. Early death was considered to be absent if the participant died on Day 101 or later, or was confirmed alive at the time of study completion/discontinuation.
Time Frame: Within 100 days or greater than 100 days after the first HSCT after the start of BESPONSA 1 mg injection up to 52 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | BESPONSA Injection 1mg (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 39
participants
  Death after HSCT in participants who underwent HSCT after starting treatment | 18
  Death within 100 days post-HSCT in participants who died after HSCT: number analyzed (Participants) | 18
  Death within 100 days post-HSCT in participants who died after HSCT | 10
  Death after > 100 days post-HSCT in participants who died after HSCT: number analyzed (Participants) | 18
  Death after > 100 days post-HSCT in participants who died after HSCT | 8
Statistical Analysis 1: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [< 18 years, ≥ 18 to < 55 years]; Test type: Other — Estimation; Risk Ratio (RR) = 0.333, 95% CI 2-sided [0.046 to 2.405] — Risk Ratio of age "< 18 years" to "≥ 18 to < 55 years"
Statistical Analysis 2: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of age [≥ 40 years, ≥ 15 to < 40 years]; Test type: Other — Estimation; Risk Ratio (RR) = 1.1, 95% CI 2-sided [0.340 to 3.560] — Risk Ratio of age "≥ 40 years" to "≥ 15 to < 40 years"
Statistical Analysis 3: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of chromosome karyotype; Test type: Other — Estimation; Risk Ratio (RR) = 1.227, 95% CI 2-sided [0.371 to 4.056] — Risk Ratio of chromosome karyotype "Philadelphia chromosome positive" to "negative"
Statistical Analysis 4: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.6, 95% CI 2-sided [0.183 to 1.966] — Risk Ratio of ECOG PS before the start of this drug "0" to "1"
Statistical Analysis 5: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of hemoglobin level immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.284 to 2.481] — Risk Ratio of hemoglobin level immediately before the start of this drug "< 10 g/dL" to "≥ 10 g/dL"
Statistical Analysis 6: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of platelet count immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 2, 95% CI 2-sided [0.604 to 6.621] — Risk Ratio of platelet count immediately before the start of this drug "< 10 × 10⁴/μL" to "≥ 10 × 10⁴/μL"
Statistical Analysis 7: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of myeloblast count immediately before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.917, 95% CI 2-sided [0.278 to 3.026] — Risk Ratio of myeloblast count immediately before the start of this drug "> 50%" to "≤ 50%"
Statistical Analysis 8: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of salvage line of the induction treatment with this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.264, 95% CI 2-sided [0.036 to 1.930] — Risk Ratio of salvage line of the induction treatment with this drug "2nd" to "1st"
Statistical Analysis 9: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of HSCT before the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 1.438, 95% CI 2-sided [0.497 to 4.161] — Risk Ratio of HSCT before the start of this drug "performed" to "not performed"
Statistical Analysis 10: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of type of the first HSCT after the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.616, 95% CI 2-sided [0.187 to 2.030] — Risk Ratio of type of the first HSCT after the start of this drug "allogeneic hematopoietic stem cell transplant with myeloablative conditioning" to "allogeneic hematopoietic stem cell transplant with nonmyeloablative conditioning"
Statistical Analysis 11: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of ECOG PS before conditioning for the first HSCT after the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 0.583, 95% CI 2-sided [0.155 to 2.192] — Risk Ratio of ECOG PS before conditioning for the first HSCT after the start of this drug "0" to "1"
Statistical Analysis 12: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of hemoglobin level before conditioning for the first HSCT after the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 2.545, 95% CI 2-sided [0.630 to 10.293] — Risk Ratio of hemoglobin level before conditioning for the first HSCT after the start of this drug "< 10 g/dL" to "≥ 10 g/dL"
Statistical Analysis 13: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of time from the date of final dose of this drug to the date of the first HSCT after the start of this drug; Test type: Other — Estimation; Risk Ratio (RR) = 1.179, 95% CI 2-sided [0.237 to 5.870] — Risk Ratio of time from the date of final dose of this drug to the date of the first HSCT after the start of this drug "≥ 4 weeks to < 8 weeks" to "< 4 weeks"
Statistical Analysis 14: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of best overall response; Test type: Other — Estimation; Risk Ratio (RR) = 2.182, 95% CI 2-sided [0.665 to 7.158] — Risk Ratio of best overall response "progression or relapse" to "complete remission (CR) or complete remission with incomplete hematologic recovery (CRi)"
Statistical Analysis 15: Comparison: BESPONSA Injection 1mg (Inotuzumab Ozogamicin); Subgroup analyses of minimal residual disease (MRD); Test type: Other — Estimation; Risk Ratio (RR) = 1.538, 95% CI 2-sided [0.392 to 6.037] — Risk Ratio of MRD "test not performed" to "negativity achieved"

11. Secondary Outcome: Hematologic Remission Rate
Description: The best overall response was evaluated for its clinical effect of hematologic remission during the observation period.
  The proportions of CR or CRi and their 95% confidence intervals were determined.
  However, if subsequent treatment for the target disease was started or HSCT was performed, the best overall response before the start of the subsequent treatment or HSCT, whichever occurred earlier, was recorded.
Time Frame: 52 Weeks. However, if subsequent treatment for the target disease was started or HSCT was performed, the best overall response before the start of the subsequent treatment or HSCT, whichever was earlier, was entered.
Population: The effectiveness analysis set excluded participants in the safety analysis set who had diseases that were outside the scope of the study. Participants without informed consent on publication of study results were excluded.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | BESPONSA Injection 1mg (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 131
Percentage | 61.8 [52.9 to 70.2]

12. Secondary Outcome: Overall Survival (OS)
Description: OS was defined and evaluated as the number of months from the start of BESPONSA Injection 1mg to all-cause death. The participant's survival status was confirmed at the time of completion or discontinuation of the study. The endpoint was censored on the day when participant's survival was last confirmed.
  For time-to-event data, the median was determined using the Kaplan-Meier method.
Time Frame: No HSCT: up to 52 weeks, HSCT: up to 104 weeks
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BESPONSA Injection 1mg (Inotuzumab Ozogamicin)
Number analyzed (Participants) | 131
Months | 10.28 [7.46 to 16.49]

ADVERSE EVENTS:
Time Frame: From first dose up to 28 days after last dose. VOD/SOS: No HSCT: up to 52 weeks, HSCT: up to 104 weeks
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | BESPONSA Injection 1mg (Inotuzumab Ozogamicin)
All-Cause Mortality (participants affected / at risk) | 21/136
Serious Adverse Events (participants affected / at risk) | 43/136
Other Adverse Events (participants affected / at risk) | 71/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BESPONSA Injection 1mg (Inotuzumab Ozogamicin) (N=136)
Aplastic anaemia (Blood and lymphatic system disorders) | 1
Cytopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 4
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 13
Bacteraemia (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Viraemia (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 4
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15
Leukaemic infiltration extramedullary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BESPONSA Injection 1mg (Inotuzumab Ozogamicin) (N=136)
Anaemia (Blood and lymphatic system disorders) | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 13
Myelosuppression (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 4
Malaise (General disorders) | 4
Pyrexia (General disorders) | 10
Hepatic function abnormal (Hepatobiliary disorders) | 4
Herpes simplex (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 9
Amylase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 5
Blood alkaline phosphatase increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 5
Hepatic enzyme increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 16
Platelet count decreased (Investigations) | 28
White blood cell count decreased (Investigations) | 9
Decreased appetite (Metabolism and nutrition disorders) | 3
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
Although this study is an all-case surveillance, the informed consent rate for disclosure of study results was 36%. It is considered that the differences observed between the results of the all-case surveillance and those obtained from patients who provided informed consent may be attributed to variations in baseline characteristics and reduced statistical precision. The main factor is presumed to be the smaller sample size, which led to wider confidence intervals and shifts in point estimates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT05923112/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT05923112/SAP_001.pdf